CLINICAL TRIAL: NCT02228590
Title: A Phase 2 Study to Examine the Safety, Tolerability and Efficacy of APL-130277 in Patients With Parkinson's Disease
Brief Title: A Study to Examine APL-130277 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTH-105
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APL-130277 (Other): open label baseline comparison
  Interventions: Drug: APL-130277

INTERVENTIONS:
Drug: APL-130277 — Apomorphine Hydrochloride, Sublingual Thin Film
  Other Names: Apomorphine Hydrochloride, Sublingual Thin Film

SUMMARY:
The primary objective of this study is to evaluate the efficacy, tolerability and safety of single treatments of APL-130277 in 16 patients with Parkinson's Disease (PD)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Clinical diagnosis of Idiopathic PD
3. Receiving stable doses of L-dopa +/- other adjunctive PD therapy for at least 4 weeks before study participation.
4. At least one OFF episode per day and a total daily OFF time of > 2 hours duration.
5. Experience predictable OFF episodes in the morning on awakening prior to receiving morning dose of levodopa.
6. Stage I to III on the Hoehn and Yahr scale in the "ON" state.
7. If female and of childbearing potential, must agree to use one of the following methods of birth control:
8. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.
9. Able to understand the consent form, and to provide written informed consent.

Exclusion Criteria:

1. Atypical or secondary parkinsonism
2. Changes in L-dopa or other PD drug dosing regimens 4 weeks before the screening visit.
3. Past treatment with any form of apomorphine within 30 days of Dosing Day 1 (patients who stopped apomorphine for reasons other than lack of efficacy OR tolerability issues may be considered for the trial).
4. Female who is pregnant or lactating.
5. Contraindications to APOKYN or hypersensitive to apomorphine hydrochloride or any of the ingredients of APOKYN (notably sodium metabisulfite), or Tigan®.
6. Participation in any other clinical trial within 14 days of the screening visit.
7. Receipt of any investigational (i.e., unapproved) medication within 30 days of the screening visit.
8. Currently taking, or likely to need to take at any time during the course of the study
9. Currently taking dopamine antagonists or depleting drugs excluding anticholinergics and/or antihistamines with anticholinergic effects.
10. Drug or alcohol dependency in the past 6 months.
11. Clinically significant orthostatic hypotension.
12. Malignant melanoma or a history of previously treated malignant melanoma within 5 years.
13. Clinically significant medical surgical or laboratory abnormality in the judgment of the investigator.
14. Psychiatric disorder, including but not limited to dementia or any disorder that, in the opinion of the Investigator requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
15. Dementia that precludes providing informed consent.
16. Potential for lack of compliance and follow-up in the judgment of the investigator.
17. Any other condition, current therapy, or prior therapy (within 30 days of the screening visit), which, in the opinion of the Investigator, would make the subject unsuitable for the study.
18. Previous neurosurgery for PD.
19. Donation of blood or plasma in the 30 days prior to dosing.
20. Presence of cankers or mouth sores.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08-31 (Actual); Primary Completion 2014-11-24 (Actual); Study Completion 2014-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (4):
- United States (4):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of South Florida Parkinson's Disease and Movement Disorders Center, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with moderate to advanced Idiopathic Parkinson's Disease (PD) were recruited to this study in 4 study sites in the United States from August 2014. The study was completed in November 2014.
Pre-assignment Details: 23 patients were screened, 20 were assigned to treatment and 1 withdrew consent prior to treatment. 19 received APL-130277
  APL-130277 sublingual film for the acute intermittent treatement of OFF episodes in PD patients
  . Doses studied were 10, 15, 20, 25 and 30 milligrams (mg).
Groups:
- APL-130277: At each dosing visit patients were assessed in a 'OFF' state by withholding their PD medication the night before, a dose of APL-130277 was administered. If the patient did not convert to a full 'ON' state within 3 hours and did not experience orthostatic hypotension, the next higher dose of APL-130277 was administered. If the patient did not turn ON with the next higher dose, levodopa was administered and completed their visit. Possible administered doses of APL-130277 were 10, 15, 20, 25 and 30 mg. Dosing Day 1: The starting dose was 10 mg APL-130277, and if no response 15 mg was administered. Dosing Day 2: Either the dose which elicited a response (i.e. an 'ON' state) at Day 1 was administered or the next higher dose (20 mg) was given. If no response occurred at 20 mg APL-130277, 25 mg was administered. Dosing Day 3: Either the dose which elicited a response at Day 2 was administered or the next higher dose (30 mg). If no response occurred at 30 mg the patient was discontinued.
Period: Overall Study
Arm/Group | APL-130277
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | APL-130277
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Resolution of an 'OFF' Episode to an 'ON' State Following Administration of APL-130277
Description: Clinical confirmation of an 'OFF' state was assessed prior to dosing and confirmation of 'OFF' or 'ON' was assessed after dosing at Visits 3 - 5 by the Investigator. The first full 'ON' dose was defined as the earliest dose in which a patient achieved a full 'ON' state as assessed by the Investigator. The percentage of patients who achieved their first full 'ON' is presented for each timepoint, regardless of the dose received, and for the study overall (i.e. all post-dose timepoints).
Time Frame: At 15, 30, 45, 60 and 90 minutes after dosing at Visits 3 - 5.
Population: The modified Intent-to-Treat (mITT) Population consisted of all patients who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | APL-130277
Number analyzed (Participants) | 19
percentage of participants
  Overall | 78.9
  15 minutes post-dose | 31.6
  30 minutes post-dose | 78.9
  45 minutes post-dose | 68.4
  60 minutes post-dose | 68.4
  90 minutes post-dose | 47.4

2. Primary Outcome: Time to 'ON' State From Time of Dosing of APL-130277
Description: Clinical confirmation of 'OFF' or 'ON' was assessed after dosing at Visits 3 - 5 by the Investigator. The time to the full 'ON' state from the time of dosing in minutes was calculated from timings noted by the Investigator and recorded in the electronic case report form (eCRF). The mean time taken for a patient to reach their first full 'ON' state following administration of APL-130277 is presented for patients who turned 'ON' for the study overall.
Time Frame: At 15, 30, 45, 60 and 90 minutes after dosing at Visits 3 - 5.
Population: The mITT Population consisted of all patients who received at least 1 dose of study medication, and data is presented for patients who turned 'ON'.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | APL-130277
Number analyzed (Participants) | 19
minutes | 24.0 (7.61)

3. Primary Outcome: Duration of 'ON' Response From Time of Dosing of APL-130277
Description: Clinical confirmation of 'OFF' or 'ON' was assessed after dosing at Visits 3 - 5 by the Investigator. The duration of the 'ON' response was defined as the length of time in which a patient was confirmed 'ON' within a dose, and was calculated from the time noted by the Investigator and recorded in the eCRF. The mean duration of the first full 'ON' response following administration of APL-130277 is presented for patients who turned 'ON' for the study overall.
Time Frame: At 15, 30, 45, 60 and 90 minutes after dosing at Visits 3 - 5.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | APL-130277
Number analyzed (Participants) | 19
minutes | 50.0 (19.36)

4. Primary Outcome: Percentage of Patients Who Completed the Trial and Experienced an 'ON' Episode
Description: Clinical confirmation of 'OFF' or 'ON' was assessed after dosing at Visits 3 - 5 by the Investigator. For the overall study, the percentage of patients who completed the trial, and who experienced an 'ON' episode is presented.
Time Frame: At 15, 30, 45, 60 and 90 minutes after dosing at Visits 3 - 5.
Population: The mITT Population consisted of all patients who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | APL-130277
Number analyzed (Participants) | 19
percentage of participants | 78.9

5. Primary Outcome: Pharmacokinetic (PK) Evaluation: Maximum Observed Plasma Concentration (Cmax)
Description: The mean Cmax values are presented for each dosage administered at Visits 3, 4, and 5 for which data was available.
  Plasma concentrations of the active substance of APL-130277, apomorphine, were analysed using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) assay, with a lower limit of quantification of 0.020 nanograms per millilitre (ng/mL).
Time Frame: Just prior to dosing and at 10, 20, 30, 45, 60 and 90 minutes after each dose at Visits 3 - 5.
Population: Blood draws for APL-130277 PK analyses were collected at select sites only. The PK Population consisted of all patients who had sufficient concentration-time data to derive noncompartmental PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | APL-130277
Number analyzed (Participants) | 8
ng/mL
  10 mg APL-130277 Dose 1 Day 1 | 2.01 (0.914)
  15 mg APL-130277 Dose 2 Day 1: number analyzed (Participants) | 6
  15 mg APL-130277 Dose 2 Day 1 | 2.52 (1.04)
  10 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 1
  10 mg APL-130277 Dose 1 Day 2 | 4.18 (NA) — No SD is available as data is for a single patient.
  20 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 7
  20 mg APL-130277 Dose 1 Day 2 | 3.82 (1.81)
  25 mg APL-130277 Dose 2 Day 2: number analyzed (Participants) | 2
  25 mg APL-130277 Dose 2 Day 2 | 4.84 (NA) — No SD available due to small number of patients analysed for this dose
  20 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 4
  20 mg APL-130277 Dose 1 Day 3 | 2.82 (1.38)
  25 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  25 mg APL-130277 Dose 1 Day 3 | 12.3 (NA) — No SD is available as data is for a single patient.
  30 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  30 mg APL-130277 Dose 1 Day 3 | 4.22 (NA) — No SD is available as data is for a single patient.
  25 mg APL-130277 Dose 2 Day 3: number analyzed (Participants) | 3
  25 mg APL-130277 Dose 2 Day 3 | 4.84 (2.99)

6. Primary Outcome: PK Evaluation: Time of Maximum Observed Plasma Concentration (Tmax)
Description: The median Tmax values are presented for each dosage administered at Visits 3, 4, and 5 for which data was available.
  Plasma concentrations of the active substance of APL-130277, apomorphine, were analysed using a validated LC-MS/MS assay, with a lower limit of quantification of 0.020 ng/mL.
Time Frame: Just prior to dosing and at 10, 20, 30, 45, 60 and 90 minutes after each dose at Visits 3 - 5.
Population: as for outcome 5
Measure: Median (Full Range); unit: minutes
Arm/Group | APL-130277
Number analyzed (Participants) | 8
minutes
  10 mg APL-130277 Dose 1 Day 1 | 60.0 [45.0 to 90.0]
  15 mg APL-130277 Dose 2 Day 1: number analyzed (Participants) | 6
  15 mg APL-130277 Dose 2 Day 1 | 35.0 [24.0 to 90.0]
  20 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 7
  20 mg APL-130277 Dose 1 Day 2 | 47.0 [25.0 to 61.0]
  20 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 4
  20 mg APL-130277 Dose 1 Day 3 | 56.5 [30.0 to 61.0]
  25 mg APL-130277 Dose 2 Day 3: number analyzed (Participants) | 3
  25 mg APL-130277 Dose 2 Day 3 | 45.0 [28.0 to 90.0]

7. Primary Outcome: PK Evaluation: Time to Last Analytically Quantifiable Concentration (Tlast)
Description: The mean Tlast values are presented for each dosage administered at Visits 3, 4, and 5 for which data was available.
  Plasma concentrations of the active substance of APL-130277, apomorphine, were analysed using a validated LC-MS/MS assay, with a lower limit of quantification of 0.020 ng/mL.
Time Frame: Just prior to dosing and at 10, 20, 30, 45, 60 and 90 minutes after each dose at Visits 3 - 5.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | APL-130277
Number analyzed (Participants) | 8
minutes
  10 mg APL-130277 Dose 1 Day 1 | 89.4 (8.63)
  15 mg APL-130277 Dose 2 Day 1: number analyzed (Participants) | 6
  15 mg APL-130277 Dose 2 Day 1 | 90.8 (2.04)
  10 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 1
  10 mg APL-130277 Dose 1 Day 2 | 95.0 (NA) — No SD is available as data is for a single patient.
  20 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 7
  20 mg APL-130277 Dose 1 Day 2 | 88.9 (15.1)
  25 mg APL-130277 Dose 2 Day 2: number analyzed (Participants) | 2
  25 mg APL-130277 Dose 2 Day 2 | 94.0 (NA) — No SD available due to small number patients analysed for this dose.
  20 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 4
  20 mg APL-130277 Dose 1 Day 3 | 95.2 (6.40)
  25 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  25 mg APL-130277 Dose 1 Day 3 | 102 (NA) — No SD is available as data is for a single patient
  30 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  30 mg APL-130277 Dose 1 Day 3 | 92.0 (NA) — No SD is available as data is for a single patient
  25 mg APL-130277 Dose 2 Day 3: number analyzed (Participants) | 3
  25 mg APL-130277 Dose 2 Day 3 | 75.7 (24.8)

8. Primary Outcome: PK Evaluation: Area Under the Plasma Concentration Time Curve, From Time 0 to 90 Minutes (AUC0-90)
Description: The mean AUC0-90 values are presented for each dosage administered at Visits 3, 4, and 5 for which data was available.
  Plasma concentrations of the active substance of APL-130277, apomorphine, were analysed using a validated LC-MS/MS assay, with a lower limit of quantification of 0.020 ng/mL.
Time Frame: Just prior to dosing and at 10, 20, 30, 45, 60 and 90 minutes after each dose at Visits 3 - 5.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | APL-130277
Number analyzed (Participants) | 8
min*ng/mL
  10 mg APL-130277 Dose 1 Day 1: number analyzed (Participants) | 7
  10 mg APL-130277 Dose 1 Day 1 | 132 (42.8)
  15 mg APL-130277 Dose 2 Day 1: number analyzed (Participants) | 6
  15 mg APL-130277 Dose 2 Day 1 | 149 (57.2)
  10 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 1
  10 mg APL-130277 Dose 1 Day 2 | 269 (NA) — No SD is available as data is for a single patient
  20 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 6
  20 mg APL-130277 Dose 1 Day 2 | 216 (127)
  25 mg APL-130277 Dose 2 Day 2: number analyzed (Participants) | 2
  25 mg APL-130277 Dose 2 Day 2 | 266 (NA) — No SD available due to small number patients analysed for this dose.
  20 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 4
  20 mg APL-130277 Dose 1 Day 3 | 170 (77.2)
  25 mg APl-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  25 mg APl-130277 Dose 1 Day 3 | 507 (NA) — No SD is available as data is for a single patient
  30 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  30 mg APL-130277 Dose 1 Day 3 | 197 (NA) — No SD is available as data is for a single patient
  25 mg APL-130277 Dose 2 Day 3: number analyzed (Participants) | 2
  25 mg APL-130277 Dose 2 Day 3 | 367 (NA) — No SD available due to small number patients analysed for this dose.

9. Primary Outcome: PK Evaluation: Area Under the Plasma Concentration Time Curve, From Time 0 to the Last Measurable Non-zero Concentration (AUClast)
Description: The mean AUClast values are presented for each dosage administered at Visits 3, 4, and 5 for which data was available.
  Plasma concentrations of the active substance of APL-130277, apomorphine, were analysed using a validated LC-MS/MS assay, with a lower limit of quantification of 0.020 ng/mL. The AUClast was calculated by a combination of linear and logarithmic trapezoidal methods (linear up/log down method).
Time Frame: Just prior to dosing and at 10, 20, 30, 45, 60 and 90 minutes after each dose at Visits 3 - 5.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | APL-130277
Number analyzed (Participants) | 8
min*ng/mL
  10 mg APL-130277 Dose 1 Day 1 | 121 (52.2)
  15 mg APL-130277 Dose 2 Day 1: number analyzed (Participants) | 6
  15 mg APL-130277 Dose 2 Day 1 | 151 (58.4)
  10 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 1
  10 mg APL-130277 Dose 1 Day 2 | 279 (NA) — No SD is available as data is for a single patient
  20 mg APL-130277 Dose 1 Day 2: number analyzed (Participants) | 7
  20 mg APL-130277 Dose 1 Day 2 | 203 (122)
  25 mg APL-130277 Dose 2 Day 2: number analyzed (Participants) | 2
  25 mg APL-130277 Dose 2 Day 2 | 277 (NA) — No SD available due to small number patients analysed for this dose.
  20 mg APL-130277 Dose 1 Day 3: number analyzed (Participants) | 4
  20 mg APL-130277 Dose 1 Day 3 | 179 (69.2)
  25 mg APl-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  25 mg APl-130277 Dose 1 Day 3 | 566 (NA) — No SD is available as data is for a single patient
  30 mg APl-130277 Dose 1 Day 3: number analyzed (Participants) | 1
  30 mg APl-130277 Dose 1 Day 3 | 206 (NA) — No SD is available as data is for a single patient
  25 mg APL-130277 Dose 2 Day 3: number analyzed (Participants) | 3
  25 mg APL-130277 Dose 2 Day 3 | 268 (193)

10. Secondary Outcome: Percentage Change in MDS-UPDRS Section III Score From Pre-dose Assessment
Description: The Motor Function section (Section III) of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms. The percent change in the MDS-UPDRS Section III score from pre-dose to the first full ON dose or last dose for non-responders is presented. A negative change from baseline indicates an improvement.
Time Frame: At 15, 30, 45, 60 and 90 minutes after dosing at Visits 3 - 5.
Population: The mITT Population consisted of all patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: percent of change
Groups:
- APL-130277: At each of 3 dosing visits patients were assessed in a practically defined 'OFF' state after withholding their usual PD medications the night before and APL-130277 sublingual film was administered initially at 10 mg. If the patient did not convert to a full 'ON' state within 3 hours from initial dosing and did not experience orthostatic
Arm/Group | APL-130277
Number analyzed (Participants) | 19
percent of change
  Change from Pre-Dose to 15 min Post-Dose | -27.9 (20.72)
  Change from Pre-Dose to 30 min Post-Dose | -34.4 (19.04)
  Change from Pre-Dose to 45 min Post-Dose | -35.6 (20.03)
  Change from Pre-Dose to 60 min Post-Dose | -32.4 (23.20)
  Change from Pre-Dose to 90 min Post-Dose | -23.8 (26.14)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were collected over a timeframe of approximately 3 months, with an onset at the time of or following the start of treatment with study medication and prior to 7 days after the end of treatment, or AEs which started prior to treatment but worsened at the time of or following the start of treatment.
Description: Adverse events are presented for the Safety Population which consisted of all patients who were enrolled into the study and received at least 1 dose of study medication.
Arm/Group | APL-130277
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (N=19)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (N=19)
nausea (Gastrointestinal disorders) | 4 (8)
vomiting (Gastrointestinal disorders) | 1 (1)
chest discomfort (General disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
muscuar weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
balance disorder (Nervous system disorders) | 1 (1)
dizziness (Nervous system disorders) | 7 (8)
headache (Nervous system disorders) | 2 (3)
paraesthesia (Nervous system disorders) | 1 (1)
somnolence (Nervous system disorders) | 6 (8)
tremor (Nervous system disorders) | 1 (2)
apathy (Psychiatric disorders) | 1 (1)
nervousness (Psychiatric disorders) | 1 (1)
yawning (Respiratory, thoracic and mediastinal disorders) | 3 (4)
upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
hot flush (Vascular disorders) | 1 (1)
orthostatic hypotension (Vascular disorders) | 1 (1)
peripheral coldness (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to the 90-minute sampling estimate λz values or calculate AUCinf, AUCext, or half-life as stated in the protocol was not possible.No PK parameters were calculated for subjects with fewer than 4 quantifiable concentrations following BLQ imputation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a mult-center publication; provided however, if a mult-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2014-09-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02228590/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02228590/SAP_001.pdf